CLINICAL TRIAL: NCT05299554
Title: A Phase 3 Open-Label Extension Study to Evaluate the Long-term Safety and Tolerability of Chronocort in the Treatment of Participants Aged 16 Years and Over With Congenital Adrenal Hyperplasia
Brief Title: Long-term Safety Study of Chronocort in the Treatment of Participants With Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-015; 2021-004467-26 (EudraCT Number)
Record Dates: First submitted 2022-01-05; First posted 2022-03-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Extension study
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Intervention Model Description: Single arm extension study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chronocort (hydrocortisone modified-release capsule) (Experimental): Chronocort (hydrocortisone modified-release capsules) supplied as 5 mg and 10 mg per capsule for oral administration.
  Interventions: Drug: Chronocort

INTERVENTIONS:
Drug: Chronocort — Hydrocortisone modified-release capsule 5 mg and 10 mg
  Other Names: Hydrocortisone modified-release hard capsule

SUMMARY:
This phase III study is an open-label extension study to be conducted at approximately 21 investigational sites across 3 countries. The study will evaluate the long-term safety and tolerability of Chronocort in participants aged 16 years and over when used as treatment for Congenital Adrenal Hyperplasia (CAH).

DETAILED DESCRIPTION:
Participants in eligible countries completing one of the specified previous Chronocort studies (DIUR-006 and DIUR 014) can either continue Chronocort treatment (if the participant received Chronocort in the feeder study) or switch to Chronocort treatment (if the participant received standard glucocorticoid therapy in the feeder study) in this open-label extension study. All participants choosing to enter this extension study will have the study procedures fully explained and informed consent obtained, prior to, or at the last visit of the feeder study. Participants who agree to take part in this extension study will then undergo the final visit of the feeder study, with the assessments conducted at the final visit also providing the baseline data for this DIUR-015 extension study where relevant (note participants who are withdrawn from treatment due to titration issues in study DIUR-014 are eligible to enter at the discretion of the Investigator, as long as all DIUR-014 safety assessments and the end of study visit are completed). Once all the baseline assessments are completed, participants will be given sufficient Chronocort to use until the next visit (the study pharmacies will be supplied with Chronocort for dispensing to participants according to the Investigators' instructions).

Outcome measures in this study will be assessed versus either the 'initial study baseline' (measurements taken at the start of participation in an interventional Chronocort study, regardless of the treatment assignment in this feeder study) or the protocol-defined 'pre-Chronocort baseline' (measurements taken prior to the first dose of continuous Chronocort) or the 'DIUR-015 baseline' (measurements taken at the start of participation in DIUR-015 study).

ELIGIBILITY:
Inclusion Criteria:

* Participants with Congenital Adrenal Hyperplasia (CAH) who have successfully completed Chronocort study DIUR-006 (sites in France and US only) or study DIUR-014.
* Participants who are capable of giving signed informed consent/assent, which includes compliance with the requirements and restrictions listed in the study's informed consent form (ICF) and in the protocol.

Exclusion Criteria:

* Participants with clinical or biochemical evidence of hepatic or renal disease e.g., creatinine >2 times the upper limit of normal (ULN) or elevated liver function tests (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >2 times the ULN).
* Participants with a history of malignancy (other than basal cell carcinoma successfully treated >26 weeks prior to entry into the study).
* Participants with a history of bilateral adrenalectomy.
* Participants with any other significant medical or psychiatric conditions that in the opinion of the Investigator would preclude participation in the study.
* Participants with a co-morbid condition requiring daily administration of a medication or consumption of any material that interferes with the metabolism of glucocorticoids.
* Participants on regular daily inhaled, topical, nasal, or oral steroids for any indication other than CAH.
* Participants anticipating regular prophylactic use of additional steroids e.g., for strenuous exercise.
* Participation in another clinical study of an investigational or licensed drug or device within 3 months prior to inclusion in this study, except for another clinical study with the current formulation of Chronocort.
* Females who are pregnant or lactating.
* Participants, who in the opinion of the Investigator, will be unable to comply with the requirements of the protocol.
* Participants who routinely work night shifts and so do not sleep during the usual night-time hours.
* Participants with a body weight of 50 kg or less (Note: this exclusion criterion is only applicable for French sites).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms of over-treatment [Safety and Tolerability] throughout the study. | Up to 32 months
  Over-replacement normally presents with chronic effects such as weight gain, increased appetite, sleeping difficulties, increased acne and Cushingoid syndrome.
Signs and symptoms of under-treatment [Safety and Tolerability] throughout the study. | Up to 32 months.
  Under-replacement normally presents with acute effects such as sudden weight loss, lack of appetite, nausea, vomiting, headache, blurred vision, fatigue, weakness, dizziness, light-headedness and syncope.
To measure signs or symptoms of under treatment [Safety and Tolerability] in terms of use of additional glucocorticoid treatment throughout the study. | Up to 32 months
  Use of Immediate Release Hydrocortisone (IRHC) from the emergency packs for stress dosing or use of any additional glucocorticoid treatment.
To measure signs or symptoms of under treatment [Safety and Tolerability] in terms of incidence of adrenal crises throughout the study. | Up to 32 months
  Occurrence of adrenal crises throughout the study.
To measure the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. | Up to 32 months
  The incidence, nature, severity, relatedness, duration, outcome, seriousness, and expectedness of treatment-emergent adverse events (TEAEs) throughout the study.
To measure the change from pre-Chronocort baseline in terms of hematology safety laboratory assessments [Safety and Tolerability]. | Up to 32 months
  Lab parameters will be summarized and compared throughout the study as follows:
  Platelet count, Red blood cell count (RBC), Haemoglobin, Haematocrit, RBC Indices: Mean corpuscular volume (MCV), Mean cell haemoglobin (MCH). Mean cell haemoglobin concentration (MCHC), Red cell distribution width (RDW).
  White blood cell (WBC) count with differential (absolute and %): Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.
To measure the change from pre-Chronocort baseline in terms of clinical chemistry safety laboratory assessments [Safety and Tolerability]. | Up to 32 months
  To measure the change from pre-Chronocort baseline in terms of clinical chemistry safety laboratory assessments [Safety and Tolerability].
  Blood urea nitrogen (BUN), Creatinine, Chloride, Total magnesium, Potassium, Sodium, Calcium, Total carbon dioxide (CO2), Inorganic phosphorus, AST/serum glutamic-oxaloacetic transaminase (SGOT), ALT/serum glutamic-pyruvic transaminase (SGPT), Alkaline phosphatase, Albumin, Total and direct bilirubin, Total protein, Lactate dehydrogenase (LDH), Total creatine kinase (CK), Uric acid.
To measure the change from pre-Chronocort baseline in terms of vital signs assessments. | Up to 32 months
  Blood pressure measurements throughout the study will be summarised and compared.

SECONDARY OUTCOMES:
To assess the impact of treatment on dose of steroid required - Change from pre-Chronocort baseline | Up to 32 months
  Change from pre-Chronocort baseline in total daily steroid dose in hydrocortisone equivalent dose at each visit.
To assess the impact of treatment on 17-Hydroxyprogesterone (17-OHP) levels - Change from pre-Chronocort baseline | Up to 32 months
  Change in 17-OHP levels from pre Chronocort baseline at each visit.
To assess the impact of treatment on Androstenedione (A4) levels - Change from pre-Chronocort baseline | Up to 32 months
  Change in A4 levels from pre-Chronocort baseline at each visit.
To assess the impact of treatment on menstrual regularity (recorded in a participant diary) as a marker of fertility - Change from pre-Chronocort baseline | Up to 32 months
  Change from pre-Chronocort baseline in menstrual regularity as recorded in a participant diary. With menstrual regularity defined as a cycle (menstrual bleeding) occurring every 21 to 35 days (only in pre-menopausal females without hysterectomy and not using hormonal contraceptives).
To assess the impact of treatment on luteinising hormone (LH) levels in men as a marker of fertility - Change from pre-Chronocort baseline | Up to 32 months
  Change from pre-Chronocort baseline in luteinising hormone (LH) levels throughout the study.
To assess the impact of treatment on testosterone by sex - Change from pre-Chronocort baseline | Up to 32 months
  Change in testosterone levels from pre-Chronocort baseline through the study, summarized by gender.
To assess the impact of treatment on waist circumference - Change from pre-Chronocort baseline | Up to 32 months
  Change from pre-Chronocort baseline to each visit in waist circumference.
To assess the impact of treatment on body weight - Change from pre-Chronocort baseline | Up to 32 months
  Change from pre-Chronocort baseline to each visit in body weight.

OTHER OUTCOMES:
To assess the impact of treatment on the dose of steroid - Change from initial study baseline daily dose | Up to 32 months
  Change from initial study baseline in daily steroid dose as the hydrocortisone equivalent dose.
To assess the impact of treatment on 17-Hydroxyprogesterone (17-OHP) levels - Change from initial study baseline | Up to 32 months
  Change in 17-OHP levels from initial study baseline throughout the study.
To assess the impact of treatment on Androstenedione (A4) levels - Change from initial study baseline | Up to 32 months
  Change in A4 levels from initial study baseline throughout the study.
To assess the impact of treatment on menstrual regularity (recorded in a participant diary) as a marker of fertility - Change from initial study baseline | Up to 32 months
  Change from initial study baseline in menstrual regularity as recorded in a participant diary. With menstrual regularity defined as a cycle (menstrual bleeding) occurring every 21 to 35 days (only in pre-menopausal females without hysterectomy and not using hormonal contraceptives).
To assess the impact of treatment on luteinising hormone (LH) levels in men as a marker of fertility - Change from initial study baseline | Up to 32 months
  Change from initial study baseline on luteinising hormone (LH) levels throughout the study.
To assess the impact of treatment on testosterone by sex - Change from initial study baseline | Up to 32 months
  Change in testosterone from initial study baseline throughout the study, summarized by gender.
To assess the impact of treatment on waist circumference - Change from initial study baseline | Up to 32 months
  Change from initial study baseline throughout the study in waist circumference.
To assess the impact of treatment on body weight - Change from initial study baseline | Up to 32 months
  Change from initial study baseline throughout the study in body weight.
To measure the change from pre-Chronocort baseline in Quality of Life (QoL) using the EuroQol 5-level Standardized Health Questionnaire (EQ 5D-5L™). | Up to 32 months
  QoL will be summarized and compared throughout the study. The scale measures on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Where the minimum score is 0 and maximum score is 100, a high score indicates a more favorable outcome.
To measure the change from initial study baseline in Quality of Life (QoL) using the EuroQol 5-level Standardized Health Questionnaire (EQ 5D-5L™). | Up to 32 months
  QoL will be summarized and compared throughout the study. The scale measures on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Where the minimum score is 0 and maximum score is 100, a high score indicates a more favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: D Merke, Principal Investigator — National Instiututes of Health Clinical Centre, Bethesda, Maryland, United States, 20892-1932
Locations (21):
- United States (11):
  - Neurocrine Investigational Site in California, Los Angeles, California
  - Neurocrine Investigational Site in California, Orange, California
  - Neurocrine Investigational Site in Florida, Jacksonville, Florida
  - Neurocrine Investigational Site in Iowa, Iowa City, Iowa
  - National Institutes of Health Center, Bethesda, Maryland
  - Neurocrine Investigational Site in Michigan, Ann Arbor, Michigan
  - Neurocrine Investigational Site in Minnesota, Rochester, Minnesota
  - Neurocrine Investigational Site in Nevada, Las Vegas, Nevada
  - Neurocrine Investigational Site in Texas, Dallas, Texas
  - Neurocrine Investigational Site in Washington, Seattle, Washington
  - Neurocrine Investigational Site in Wisconsin, Milwaukee, Wisconsin
- France (6):
  - Neurocrine Investigational Site in Caen, Caen
  - Neurocrine investigational Site in Lyon, Lyon
  - Neurocrine Investigational Site in Paris, Paris
  - Neurocrine Investigational Site in Pessac, Pessac
  - Neurocrine Investigational Site in Toulouse (Children's hospital), Toulouse
  - Neurocrine Investigational Site in Toulouse, Toulouse
- Japan (4):
  - Neurocrine Investigational Site in Asahi-ku, Yokohama, Kanagawa
  - Neurocrine Investigational Site in Yushima, Bunkyō-Ku, Tokyo
  - Neurocrine Investigational Site in Okura, Setagaya-Ku, Tokyo
  - Neurocrine Investigational Site in Toyama, Shinjuku-Ku, Tokyo